CLINICAL TRIAL: NCT05282563
Title: A Multicenter, Open, Single Arm Clinical Study on the Safety of Double and a Half Layered Esophagojejunal Anastomosis in Curative Gastrectomy
Brief Title: Clinical Study on the Safety of Double and a Half Layered Esophagojejunal Anastomosis in Curative Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Luoyang Central Hospital (Other); Nanyang Central Hospital (Other); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Kaifeng Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAFT
Record Dates: First submitted 2021-11-29; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2021-05

CONDITIONS: Surgery--Complications
Keywords: Gastricneoplasms; gastrectomy; Esophagojejunal anastomosis; Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The safety of esophagojejunostomy in total gastrectomy for gastric cancer (Other): The safety of esophagojejunostomy depends on the integrity of the anastomosis, sufficient blood supply and satisfactory tension. Early tight mucosal anastomosis and the proliferation of mucosal epithelial cells can reduce the stimulation of digestive fluid to the anastomotic wound.Professor Zhao Yuzhou surgical team proposed double and a half layered esophagojejunal anastomosis to improve the safety of anastomosis. This method is simple and has no special requirements for the selection of instruments and sutures. It can be carried out in all levels of hospitals. In order to verify the value of this method in gastrointestinal reconstruction of gastric cancer, Professor Zhao Yuzhou surgical team plans to carry out a multicenter, randomized controlled study throughout the province.
  Interventions: Procedure: double and a half layered esophagojejunal anastomosis

INTERVENTIONS:
Procedure: double and a half layered esophagojejunal anastomosis — After the end of esophagojejunostomy, 3/0 barbed suture or absorbable suture was used. First, the anastomotic site was sutured continuously for one circle, with the suture spacing of 3-4 mm and the width of 4-5 mm. Then, the continuous horizontal mattress type seromuscular layer varus suture was used to embed the anastomotic stoma for one circle, and the suture width was 5~8 mm above and below the anastomotic stoma. After the completion of esophagojejunostomy, the full-thickness reinforcement of the anastomosis and the embedding of the seromuscular layer can ensure the complete anastomosis of the mucosal layer of the anastomosis. The embedding of the seromuscular layer can also improve the anti-pressure and anti-tension of the anastomosis, and provide a guarantee for the primary healing of the anastomosis.

SUMMARY:
Surgical resection remain the main means for gastric cancer. With the improvement of surgical techniques and concepts, the incidence of postoperative complications gradually decreased, but esophagojejunostomy complications occur frequently. Studies have showed that the risks of esophagojejunostomy leakage related to old age, obesity, malnutrition, neoadjuvant radiotherapy and chemotherapy, and the incidence rate was 1%-16.5%. The incidence of anastomotic leakage varies greatly, which suggests that effective preventive measures can reduce the probability of anastomotic leakage. In addition to the patient factors, the technique and experience of the operator are also important to reduce anastomotic leakage.

The safety of esophagojejunostomy depends on the integrity of the anastomosis, sufficient blood supply and satisfactory tension. Early tight mucosal anastomosis and the proliferation of mucosal epithelial cells can reduce the stimulation of digestive fluid to the anastomotic wound. However, there are some problems in the operation: 1. When esophagojejunostomy is completed with tubular stapler, it is the contraposition of the plasma muscular layer of the digestive tract; 2. Because of the different diameter of esophagojejunostomy and tissue hypertrophy, the internal mucosa layer of the anastomosis is often torn or the residual tissue is embedded in the anastomosis, which affects the healing of the anastomosis.

Double and a half layered esophagojejunal anastomosis was proposed to improve the safety of anastomosis. The procedure is as follows: after the end of esophagojejunostomy, 3/0 barbed suture or absorbable suture was used. First, the anastomotic site was sutured continuously for one circle, with the suture spacing of 3-4 mm and the width of 4-5 mm. Then, the continuous horizontal mattress type seromuscular layer varus suture was used to embed the anastomotic stoma for one circle, and the suture width was 5-8 mm above and below the anastomotic stoma. After the completion of esophagojejunostomy, the full-thickness reinforcement of the anastomosis and the embedding of the seromuscular layer can ensure the complete anastomosis of the mucosal layer of the anastomosis. The embedding of the seromuscular layer can also improve the anti-pressure and anti-tension of the anastomosis, and provide a guarantee for the primary healing of the anastomosis.

DETAILED DESCRIPTION:
Surgical resection remain the main means for gastric cancer. How to reconstruct the digestive tract after total gastrectomy for gastric cancer is a hot topic for clinicians. Compared to jejunojejunostomy, esophagojejunostomy is difficult to operate. With the development of endoscopic technique, more and more methods of total laparoscopic esophagojejunostomy have been developed in clinic and accepted by surgeons. However, due to the requirements of laparoscopic surgery for gastric cancer staging and the high cost of total laparoscopic digestive tract reconstruction, most doctors still choose open surgery or laparoscopic assisted radical gastrectomy. Esophagojejunostomy is the main method for digestive tract reconstruction.

With the improvement of surgical techniques and concepts, the incidence of postoperative complications gradually decreased, but esophagojejunostomy complications occur frequently. Studies have showed that the risks of esophagojejunostomy leakage related to old age, obesity, malnutrition, neoadjuvant radiotherapy and chemotherapy, and the incidence rate was 1%-16.5%. The incidence of anastomotic leakage varies greatly, which also suggests that effective preventive measures can reduce the probability of anastomotic leakage. In addition to the patient factors, the technique and experience of the operator are also important to reduce anastomotic leakage. For esophagojejunostomy in surgery, most doctors believe that simple instrument anastomosis can not avoid the occurrence of anastomotic leakage, and need to strengthen the anastomotic. At the same time, anastomotic reinforcement can not completely avoid the occurrence of anastomotic leakage.

The safety of esophagojejunostomy depends on the integrity of the anastomosis, sufficient blood supply and satisfactory tension. Early tight mucosal anastomosis and the proliferation of mucosal epithelial cells can reduce the stimulation of digestive fluid to the anastomotic wound. However, there are some problems in the operation: 1. When esophagojejunostomy is completed with tubular stapler, it is the contraposition of the plasma muscular layer of the digestive tract; 2. Because of the different diameter of esophagojejunostomy and tissue hypertrophy, the internal mucosa layer of the anastomosis is often torn or the residual tissue is embedded in the anastomosis, which affects the healing of the anastomosis.

Professor Zhao Yuzhou surgical team proposed double and a half layered esophagojejunal anastomosis to improve the safety of anastomosis. The procedure is as follows: after the end of esophagojejunostomy, 3/0 barbed suture or absorbable suture was used. First, the anastomotic site was sutured continuously for one circle, with the suture spacing of 3-4 mm and the width of 4-5 mm. Then, the continuous horizontal mattress type seromuscular layer varus suture was used to embed the anastomotic stoma for one circle, and the suture width was 5-8 mm above and below the anastomotic stoma. After the completion of esophagojejunostomy, the full-thickness reinforcement of the anastomosis and the embedding of the seromuscular layer can ensure the complete anastomosis of the mucosal layer of the anastomosis. The embedding of the seromuscular layer can also improve the anti-pressure and anti-tension of the anastomosis, and provide a guarantee for the primary healing of the anastomosis.

This method is simple and has no special requirements for the selection of instruments and sutures. It can be carried out in all levels of hospitals. It should be noted that simple improvement of anastomosis can not completely eliminate anastomotic complications, but still need to cooperate with surgical drainage, nutritional support and other measures to reduce the harm of postoperative anastomotic leakage. Professor Zhao Yuzhou surgical team used this method to complete more than 800 gastric cancer operations. The results showed that double and a half layered esophagojejunal anastomosis can significantly reduce the incidence of anastomotic leakage and prevent anastomotic bleeding, and without increasing the incidence of anastomotic stenosis. The results have been published in chinese Journal of gastrointestinal surgery.

In order to further verify the value of this method in gastrointestinal reconstruction of gastric cancer,Professor Zhao Yuzhou surgical team plans to carry out a multicenter, randomized controlled study throughout the province.

ELIGIBILITY:
Inclusion Criteria:

1. The patients voluntarily participated in the study and signed the informed consent
2. 18 years old≤75 years old
3. The primary gastric lesion was diagnosed as gastric adenocarcinoma by endoscopic biopsy
4. Patients scheduled for radical gastrectomy with esophagojejunostomy (also applicable for multiple primary cancers)
5. ECOG physical status score 0/1
6. ASA score I-III
7. The expected survival time is more than 12 weeks
8. The patient agreed to accept the operation and signed the informed consent form to undertake the risk of the operation

Exclusion Criteria:

1. Other malignant tumors occurred or coexisted within 5 years
2. History of upper abdominal surgery (except laparoscopic cholecystectomy)
3. History of gastric surgery (except for patients who failed ESD/EMR for gastric cancer and needed radical gastrectomy and planned esophagojejunostomy)
4. Pregnant or lactating women
5. Have a history of psychotropic drug abuse and can not quit or have mental disorders
6. Patients with severe cachexia, inability to eat or tolerate surgery
7. Preoperative imaging examination showed that the tumor invaded the surrounding organs and regional fusion enlarged lymph nodes (maximum diameter≥3cm) and could not be radical resection
8. A history of unstable angina or myocardial infarction within 6 months There was a history of cerebral infarction or cerebral hemorrhage within 6 months
9. There was a history of continuous systemic corticosteroid therapy within 1 month
10. Other diseases need to be treated by surgery at the same time
11. Gastric cancer complications (bleeding, perforation, obstruction) need emergency surgery
12. Pulmonary function test FEV1<50% of predicted value
13. Patients with any severe and/or uncontrolled disease include:

    1. Patients with hypertension who can not be well controlled by antihypertensive drugs (systolic blood pressure≥150 mmHg, diastolic blood pressure≥100 mmHg);
    2. Patients with grade I or above myocardial ischemia or myocardial infarction, arrhythmia (including QTc≥480ms) and grade 2 or above congestive heart failure (NYHA classification);
    3. Active or uncontrolled severe infection (≥CTCAE grade 2 infection);
    4. Renal failure requires hemodialysis or peritoneal dialysis;
    5. History of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or organ transplantation;
    6. The patients with poor glycemic control (FBG>10mmol/L);
    7. Patients with epilepsy and need treatment;
14. According to the judgment of the researchers, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of complications after the operation | 1 months
  Criteria for determining complications: all postoperative complications were graded by Clavien⁃Dindo grading system. Complications of grade III and above were defined as serious complications.Judgment of anastomotic complications: (1) anastomotic leakage (2) Anastomotic bleeding (3) Anastomotic stenosis.
The incidence of operative mortality after the operation | 1 months
  Death after the operation

SECONDARY OUTCOMES:
Long term complications | One year later
  Criteria for determining complications: all postoperative complications were graded by Clavien⁃Dindo grading system. Complications of grade III and above were defined as serious complications.Judgment of anastomotic complications: (1) anastomotic recurrence (2) Anastomotic stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Li Sen, Dr, Study Director — Affiliated Cancer Hospital of Zhengzhou University
Locations (1):
- Henan cancer hopital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma PF, Cao YH, Zhang JL, Liu CY, Zhang XJ, Li S, Han GS, Zhao YZ. [Safety of two and a half layered esophagojejunal anastomosis in total gastrectomy for gastric cancer]. Zhonghua Wei Chang Wai Ke Za Zhi. 2020 Oct 25;23(10):969-975. doi: 10.3760/cma.j.cn.441530-20191010-00445. Chinese. PMID 33053992
- [Background] Sun Y, Fang Y. [Prevention and treatment of anastomosis complications after radical gastrectomy]. Zhonghua Wei Chang Wai Ke Za Zhi. 2017 Feb 25;20(2):144-147. Chinese. PMID 28226346
- [Background] Takeuchi D, Koide N, Suzuki A, Ishizone S, Shimizu F, Tsuchiya T, Kumeda S, Miyagawa S. Postoperative complications in elderly patients with gastric cancer. J Surg Res. 2015 Oct;198(2):317-26. doi: 10.1016/j.jss.2015.03.095. Epub 2015 Apr 4. PMID 26033612
- [Background] Li HZ, Liu ZY, Ahmed A, Fu HQ. [Comparative observation of microcirculation and tissue healing process in gastrointestinal anastomosis with apposition or inverted suturing]. Zhonghua Wei Chang Wai Ke Za Zhi. 2011 Jan;14(1):57-60. Chinese. PMID 21271383
- [Background] Wang GC, Liu YJ, Cheng Y, Wang YC, Liu XY, Han GS. [Prevention of high-risk complications for high esophagojejunal anastomosis leakage after total gastrectomy]. Zhonghua Zhong Liu Za Zhi. 2017 Oct 23;39(10):792-794. doi: 10.3760/cma.j.issn.0253-3766.2017.10.014. No abstract available. Chinese. PMID 29061026
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Ren JA, Li JS. [Early diagnosis and rapid treatments of gastrointestinal fistula]. Zhonghua Wei Chang Wai Ke Za Zhi. 2006 Jul;9(4):279-80. Chinese. PMID 16886101